CLINICAL TRIAL: NCT05144191
Title: Insignia™ Hip Stem Outcomes Study - A Prospective, Post-market, Multi-center Evaluation of the Clinical Outcomes of the Insignia™ Hip Stem for Total Hip Replacement Surgery
Brief Title: Insignia™ Hip Stem Outcomes Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 107
Record Dates: First submitted 2021-11-03; First posted 2021-12-03 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Hip Osteoarthritis; Avascular Necrosis; Rheumatoid Arthritis; Post-traumatic Osteoarthritis; Femoral Neck Fractures; Trochanteric Fractures; Surgery
MeSH Terms: conditions — Osteoarthritis, Hip; Osteonecrosis; Arthritis, Rheumatoid; Femoral Neck Fractures; Hip Fractures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Insignia uncemented Hip Stem (Other): The Insignia™ Hip Stem is a collared stem that features a plasma-sprayed Hydroxyapatite (HA) coating over plasma-sprayed titanium in the proximal region and a plasma-sprayed HA coating over grit blast in the distal region and collar underside.
  Insignia™ Hip Stems are intended for 'cement less' use only and are intended for total arthroplasty procedures.
  Interventions: Device: Insignia uncemented Hip Stem

INTERVENTIONS:
Device: Insignia uncemented Hip Stem — Device: Replacement of arthritic hip with Insignia uncemented Hip Stem

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of the Insignia™ Hip Stem for global market access and post-market clinical follow-up up to 10 years postoperative.

DETAILED DESCRIPTION:
This study is a prospective, post-market, multi-center clinical investigation of the Insignia™ Hip Stem for primary and revision total hip arthroplasty (THA) in a consecutive series of patients who meet the eligibility criteria. The total enrollment goal for the study is a minimum of 313 cases, all of which will receive the Insignia™ Hip Stem.

ELIGIBILITY:
Inclusion Criteria:

* The subject has signed an Institutional Review Board (IRB)-approved, study specific Informed Consent Form (ICF).
* The subject is skeletally mature
* The subject has a diagnosis as listed in the instructions for use (IFU), which include non inflammatory degenerative joint disease (including osteoarthritis or avascular necrosis), rheumatoid arthritis or post-traumatic arthritis, correction of functional deformity, treatment of nonunion, femoral neck and trochanteric fractures.
* The subject is a candidate for a primary or revision cementless THA.
* The subject is willing and able to comply with postoperative scheduled clinical evaluations.

Exclusion Criteria:

* The subject is pregnant or breastfeeding
* The subject has an active or suspected latent infection in or about the affected hip joint at the time of study device implantation.
* The subject has any mental or neuromuscular disorder which would create an unacceptable risk of prosthesis instability, prosthesis fixation failure, or complications in postoperative care.
* The subject has bone stock compromised by disease, infection or prior implantation which cannot provide adequate support and/or fixation to the prosthesis.
* The subject is immunologically suppressed or receiving steroids in excess of normal physiological requirements (e.g. > 30 days).
* The subject has a known sensitivity to device materials.
* The subject is involved in any ongoing legal matter, investigation, or dispute pertaining to the operative site.
* The subject is a prisoner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2034-04-02 (Estimated); Study Completion 2034-04-02 (Estimated)

PRIMARY OUTCOMES:
Survival Rate | 10 years
  Evaluation of the survival rate for Insignia Hip Stem is defined as absence of femoral stem revision for aseptic loosening or device-related femoral fracture.
Harris Hip Score (HHS) | 10 Years
  The Harris Hip Score (HHS) assesses pain, function, joint deformity and range of motion.
  Scores can range from 0 to 100 with 0 being the worst and 100 being the best score.
  A score of 80-100 is considered good-excellent and a score of less than or equal to 79 is considered fair-poor. 90-100 = excellent 80-89 = good 70-79 = fair 0-69 = poor

SECONDARY OUTCOMES:
Harris Hip Score (HHS) | pre-op, 6 week, 1,2,5 and 7 years
  The Harris Hip Score (HHS) assesses pain, function, joint deformity and range of motion.
  Scores can range from 0 to 100 with 0 being the worst and 100 being the best score.
  A score of 80-100 is considered good-excellent and a score of less than or equal to 79 is considered fair-poor. 90-100 = excellent 80-89 = good 70-79 = fair 0-69 = poor
EQ-5D - Descriptive System | pre-op, 6 week, 1,2,3, 4,5,7 and 10 years
  The EuroQol-5 Dimension (EQ-5D) is a subject-completed questionnaire designed to assess subject health state values.
  The EQ-5D descriptive system comprises the following five dimensions: mobility self care, usual activities, pain/comfort and anxiety/depression. Each dimension has 3 levels indicating no problems, some problems or extreme problems. The index values on a scale between -1 (low) and 1 (high) are showing the average health status according to the 5 dimensions: A low score shows worse health and a high score shows better health.
EQ-5D - Visual analogue scale (VAS) | pre-op, 6 week, 1,2,3, 4,5,7 and 10 years
  The EuroQol-5 Dimension (EQ-5D) is a subject-completed questionnaire designed to assess subject health state values.
  With the EQ Visual Analogue Scale (VAS) the respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).
Survival Rate | 2 years
  Evaluation of the survival rate for Insignia™ Hip Stem is defined as absence of femoral stem revision for aseptic loosening or device-related femoral fracture
  Success rate at two (2) years postoperative with the Insignia™ Hip Stem is not worse than 98 % with a non-inferiority margin of 3.5%.
  Success rate at 10 years postoperative with the Insignia™ Hip Stem is not worse than 95% with a non-inferiority margin of 5%.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - The MORE Foundation, Phoenix, Arizona
  - University of California, San Francisco, San Francisco, California
  - Midwest Orthopaedics at Rush, Chicago, Illinois
  - Reno Orthopedic Center Foundation, Reno, Nevada
  - Northwell Health: University Orthopaedic Associates, Great Neck, New York
  - OrthoCarolina Research Institute, Charlotte, North Carolina
  - Alleghany Health Network- Research Institute, Pittsburgh, Pennsylvania
  - TOA Research Foundation, Nashville, Tennessee
  - Baylor Scott and White Medical Center, Temple, Texas
  - Orthopedic Physician Associates, Seattle, Washington
  - Providence Orthopedics and Sports Medicine, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No